CLINICAL TRIAL: NCT01612286
Title: A Phase II Clinical Study of Endostar Combination With Chemotherapy in the Metastatic Nasopharyngeal Carcinoma
Brief Title: Endostar Combination With Chemotherapy for the Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhejaingCH-npc-02
Record Dates: First submitted 2012-05-28; First posted 2012-06-05 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2013-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Recombinant human endostatin; nasopharyngeal carcinoma; chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Endostatins; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- endostatin (Experimental): chemotherapy concurrently with endostatin
  Interventions: Drug: endostatin

INTERVENTIONS:
Drug: endostatin — Gemcitabine 1.0g/m2 d1,8 cisplatin 80mg/m2 endostatin 15mg/d 14days/cycle *4cycles
  Other Names: endostar

SUMMARY:
The investigators designed this study to evaluate the efficiency and the acute toxicities of recombinant human endostatin (endostar) combined with chemotherapy in the metastatic nasopharyngeal carcinoma (NPC).

DETAILED DESCRIPTION:
To evaluate the progression free survival (PFS), overall survival (OS), Acute adverse reaction of recombinant human endostatin (endostar) combined with chemotherapy to the metastatic nasopharyngeal carcinoma (NPC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed metastatic NPC patient who have received radiotherapy or chemoradiotherapy with an at least 6 months interval
* Have measurable lesions
* No dysfunction of the major organs
* Can understand this study and give a signed informed consent certificates
* without a history of allergic reaction to the biological agents

Exclusion Criteria:

* Pregnant or lactating women; Women of child-bearing age without contraception
* with a Serious infection or dysfunction of the major organs
* have taken other antitumor drugs during the period of 30 days ahead of this clinical trial
* allergic to the Escherichia coli preparations
* Cann't understand this study and give a signed informed consent certificates

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
progress free survival(PFS) | 1 year and 2years
  PFS means assignament to the date of any local or distant progress of the disease useing Kaplan-Meier caculate the progress free survival rates

SECONDARY OUTCOMES:
overall survival(OS) | baseline to date of death from any cause
  the overall survival denote to assignment to date of death from any cause. Using Kaplan-Meier to caculate the 1-year ,2-year,3-year overall survival rate
Adverse events | participants will be followed for the duration of hospital stay,an expected average of 100 days and every 3 months thereafter for 1 year
  observe and record the toxicity profile(incluing but not limit to mocositis,liver and kidney function,et al.)according NCI-CTCAE(3rd edtion) during the chemotherapy,Targeted therapy and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bin Li, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang cancer hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Jin T, Li B, Chen XZ. A phase II trial of Endostar combined with gemcitabine and cisplatin chemotherapy in patients with metastatic nasopharyngeal carcinoma (NCT01612286). Oncol Res. 2013;21(6):317-23. doi: 10.3727/096504014X13983417587401. PMID 25198661